CLINICAL TRIAL: NCT03812133
Title: Risk Factors and Reasons for Cancellation Within 24 Hours of Scheduled Elective Surgery in an Academic Medical Centre
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-2286
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Operating Theatre Cancellations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical patients: Patients who were electively scheduled for surgery.

SUMMARY:
The Operating Theatre (OT) is the largest cost centre as well as the main revenue generator in most hospitals. One of the common problems affecting optimal OT utilization is the cancellation of scheduled surgeries. The goal of this study was to identify factors associated with cancellation within 24 hours of scheduled surgeries in a tertiary hospital

DETAILED DESCRIPTION:
The Operating Theatre (OT) is the largest cost centre as well as the main revenue generator in most hospitals. The operating theatre involves significant resources - materials, medications and manpower. One of the common problems affecting optimal OT utilization is the cancellation of scheduled surgeries. This results in a significant waste of resources, especially when cancellation occurs within 24 hours of the scheduled surgery, when it is too late to arrange replacement surgery. Cancellation also impacts the patient and their families.

Reported cancellation rates range between 5% to 40%. Reasons for cancellations vary, including patient factors, surgeon factors, and system issues relating to the preoperative anaesthesia assessment clinic attendance, the surgery itself, and the availability of post-surgical care facilities. Between 60% to 90% of cancellations have been reported to be potentially avoidable.

The goal of this study was to identify factors associated with cancellation within 24 hours of scheduled surgery in a tertiary academic hospital, and the reasons for cancellation, with the goal of identifying areas for intervention to reduce avoidable surgery cancellations and reduce unnecessary waste.

ELIGIBILITY:
Adult patients (age 18 years and older) who were scheduled for elective surgery at the Singapore General Hospital main operating theatre or ambulatory surgical centre, regardless of surgical discipline, or residency, were included in the study. Only the first surgery in the study period was included if a patient had multiple surgeries over this period. Minor surgeries under local anaesthesia were also excluded. We excluded those without previous admissions in the past 3 years prior to the surgery, as data for chronic disease history and healthcare utilization patterns were not available for these patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The median patient age was 68 years (IQR 63 - 75 years), with 44% being male patients and 80% Chinese. Majority were Singapore citizens or permanent residents (98%). Two-thirds of the surgical patients were in a subsidized ward class (2665, 66%). Only 2% required Medifund assistance.
Sampling Method: Non-Probability Sample
Enrollment: 4060 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Cancellation | 24 hours of surgery
  Cancellation of surgery within 24 hours of procedure